CLINICAL TRIAL: NCT06594211
Title: A Single-Arm, Open-Label Study of Allogeneic Anti-BCMA/GPRC5D Bispecific CAR-NK Cells (ACT-001) in Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: Allogeneic Anti-BCMA/GPRC5D Bispecific CAR-NK Cells (ACT-001) in Patients With Relapsed or Refractorymultiple Myeloma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Collaborators: Acellytron Therapeutics (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LYC2024-007
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ACT-001 CAR-NK cell (Experimental)
  Interventions: Biological: ACT-001 CAR-NK cell

INTERVENTIONS:
Biological: ACT-001 CAR-NK cell — Subjects were distributed into three dosage groups, each receiving a single dose of CAR-NK cells at levels of 1×10^8, 3×10^8, and 9×10^8 cells, respectively.

SUMMARY:
This is a single-arm, open-label, exploratory clinical study to evaluate the safety and efficacy of allogeneic anti-BCMA/GPRC5D bispecific chimeric antigen receptor natural killer (CAR-NK) cells (ACT-001) in patients with refractory or relapsed multiple myeloma (r/r MM).

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 to 75 years inclusive, with no gender restrictions.
2. Expected survival time exceeding 12 weeks.
3. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-2.
4. Documented diagnosis of relapsed or refractory multiple myeloma (RRMM), and meets the following conditions:

   * Relapsed or refractory after at least three prior lines of therapy, including proteasome inhibitors, immunomodulatory agents, and anti-CD38 monoclonal antibodies, with at least one complete cycle of treatment for each line, unless progressive disease (PD) was documented as the best response to that line.
   * Disease progression during the most recent treatment or within 12 months.
5. Measurable disease at screening as defined by at least one of the following:

   * Serum M protein ≥ 5 g/L.
   * Urine M protein ≥ 200 mg/24h.
   * Involved serum free light chain ≥ 100 mg/L and abnormal serum free light chain κ/λ ratio.
6. Oxygen saturation ≥ 95% within 3 days prior to cell infusion.
7. Clinical laboratory values meeting the following criteria at screening:

   * Hemoglobin ≥ 80 g/L (without red blood cell transfusion within 7 days prior to testing; use of recombinant human erythropoietin is allowed).
   * Platelet count ≥ 50 × 10^9/L (without platelet transfusion or treatment with recombinant human thrombopoietin or thrombopoietin receptor agonists within 7 days prior to testing).
   * Absolute neutrophil count (ANC) ≥ 0.75 × 10^9/L (use of growth factors is allowed, but not within 7 days prior to testing).
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3.0 × upper limit of normal (ULN).
   * Creatinine clearance ≥ 40 mL/min, calculated based on the Cockcroft-Gault formula.
   * Total bilirubin ≤ 2.0 × ULN; for participants with congenital bilirubin encephalopathy (such as Gilbert's syndrome), direct bilirubin must be ≤ 1.5 × ULN.
   * Corrected serum calcium ≤ 12.5 mg/dL (≤ 3.1 mmol/L) or ionized calcium ≤ 6.5 mg/dL (≤ 1.6 mmol/L).
   * For participants who meet the inclusion criteria at screening, red blood cell transfusion may be performed as needed after screening to maintain hemoglobin levels ≥ 80 g/L.
8. Deemed by the investigator to be able to receive lymphocyte-depleting chemotherapy.
9. Male participants and females of childbearing potential must agree to use effective contraception from the time of signing the Informed Consent Form (ICF) until 2 years after receiving the study drug. Females of childbearing potential must have a negative serum pregnancy test prior to receiving the study drug.
10. The participant can understand the study and has signed the ICF.
11. Participants who have previously received BCMA or GPRC5D targeted therapy, including but not limited to CAR-T, antibody-drug conjugates (ADCs), or bispecific antibodies, are allowed to participate in the study.

Exclusion Criteria:

1. Pregnant or breastfeeding women; and subjects planning pregnancy within 2 years after signing the Informed Consent Form (ICF) until after receiving the study medication.
2. Presence of uncontrollable active infections requiring parenteral antibacterials, antivirals, or antifungals; positivity for Hepatitis B surface antigen (HbsAg) or Hepatitis B core antibody (HbcAb), with detectable Hepatitis B Virus (HBV) DNA in peripheral blood; positivity for Hepatitis C Virus (HCV) antibody and HCV RNA in peripheral blood; positivity for TRUST test for syphilis; positivity for Human Immunodeficiency Virus (HIV) antibody.
3. Subjects deemed by the investigator to have significant dysfunction of vital organs (cardiovascular, pulmonary); subjects with gastrointestinal active bleeding within 3 months prior to signing the ICF; uncontrolled hypertension (systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 95 mmHg), hypertensive crisis, or history of hypertensive encephalopathy; history or evidence of significant cardiovascular or cerebrovascular risk, including congestive heart failure (New York Heart Association class ≥ III), left ventricular ejection fraction < 50%, unstable angina, clinically significant arrhythmias (such as ventricular fibrillation, ventricular tachycardia, etc.); history of arterial thrombosis (such as stroke, transient ischemic attack) within 3 months prior to signing the ICF; history of symptomatic deep vein thrombosis, pulmonary embolism within 6 months prior to signing the ICF, or history of coronary artery angioplasty, defibrillation, or any clinical complications or diseases that may pose risks to the subject's safety or interfere with the study evaluation, procedures, or completion.
4. History or current evidence of any condition or disease that could interfere with the study results or, in the opinion of the investigator, is not in the best interest of the patient to participate.
5. Active central nervous system disease, or a history of the central nervous system requiring treatment (such as epilepsy); or subjects with central nervous system metastatic disease, leptomeningeal disease, or metastatic spinal cord compression.
6. Systemic corticosteroid therapy within 1 week prior to treatment, excluding the following: intranasal, inhaled, or local corticosteroids, local corticosteroid injections (such as intra-articular injections), systemic corticosteroid therapy at a daily dose not exceeding 10 mg of prednisone or its equivalent physiological dose, and corticosteroids used as premedication for allergic reactions.
7. Prior antitumor therapy as follows, within the specified time frames prior to cell infusion: (a) Targeted therapy, proteasome inhibitors, or cytotoxic therapy within 2 weeks; (b) Immunomodulatory agent therapy within 1 week; (c) Monoclonal antibody treatment for multiple myeloma within 3 weeks; (d) Radiotherapy within 2 weeks. However, subjects are eligible irrespective of the end date of radiotherapy if the radiation field covered ≤ 5% of the bone marrow reserve.
8. Prior therapy with any other investigational drugs or systemic anticancer treatments within 4 weeks prior to signing the ICF.
9. History of another primary malignancy within 3 years prior to starting the study treatment, with exceptions for the disease under study, adequately treated basal or squamous cell carcinoma of the skin, and in situ cervical cancer.
10. Subjects with a history or presence of interstitial lung disease or interstitial pneumonia.
11. Subjects planning to undergo autologous stem cell transplantation (ASCT) during the study.
12. Known hypersensitivity to any component of the anti-human BCMA×GPRC5D CAR-NK cell injection or the lymphodepletion regimen (cyclophosphamide and fludarabine).
13. Subjects who have undergone major surgery within 2 weeks or received live attenuated vaccines within 4 weeks prior to the pretreatment regimen.
14. Any investigator-assessed complications or other conditions that may affect a subject's ability to comply with the protocol or make them unsuitable to participate in the study.
15. Subjects with mental disorder who are unable to provide written ICF or comply with study procedures; or those unwilling or unable to adhere to study requirements.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-10-09 (Estimated); Primary Completion 2028-10-09 (Estimated); Study Completion 2028-10-09 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | From admission to 28 days after CAR-NK cells infusion
  Adverse events assessed according to NCI-CTCAE v5.0 criteria
Incidence and type of adverse events (AEs) | From admission to 2 years after CAR-NK cells infusion
  To identify the incidence and the type of AEs, including abnormalities in clinical, laboratory assessments, ECGs, echocardiography, vital sign assessments, and physical exams.

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China